CLINICAL TRIAL: NCT01289314
Title: A Comparison of Long Term Outcomes Following Total Laparoscopic Hysterectomy and Laparoscopic Supracervical Hysterectomy.
Brief Title: Long Term Outcomes Following Total Laparoscopic Hysterectomy and Laparoscopic Supracervical Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Espen Berner / Marit Lieng, Dept. of Gynecology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAP-HYST-TRIAL
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Total Laparoscopic Hysterectomy; Laparoscopic Supracervical Hysterectomy; Fibromas; Abnormal Uterine Bleeding; Dysmenorrhea
Keywords: total laparoscopic hysterectomy; laparoscopic supracervical hysterectomy
MeSH Terms: conditions — Fibroma; Metrorrhagia; Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total laparoscopic hysterectomy (Active Comparator)
  Interventions: Procedure: TLH
- Laparoscopic supracervical hysterectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic supracervical hysterectomy

INTERVENTIONS:
Procedure: TLH — Total laparoscopic hysterectomy (TLH)
  Arms: Total laparoscopic hysterectomy
Procedure: Laparoscopic supracervical hysterectomy — Laparoscopic supracervical hysterectomy (LSH)
  Arms: Laparoscopic supracervical hysterectomy

SUMMARY:
Objective: To compare the occurrence and intensity of pelvic pain as well as patient satisfaction and quality of life after total laparoscopic and laparoscopic supracervical hysterectomy.

Design: Prospective randomised trial.

Null hypothesis 1: There is no significant difference in occurrence and intensity of pelvic pain following TLH compared with following LSH.

Null hypothesis 2: There is no significant difference in patient satisfaction and quality of life following TLH compared with following LSH.

DETAILED DESCRIPTION:
Sample: 62 consecutive premenopausal women referred to the department for hysterectomy on the basis of a benign condition. The expected mean pain reduction (m) in the LSH group: 3.32, sd (s): 2.71.24 A difference in mean pain reduction (d) equal to 1 sd is considered a clinically important improvement (standardised difference d/s=1). Number of women required (power 90 % and a level of significance 0.05): 62 patients.

Methods: The study participants are randomised to total laparoscopic hysterectomy (n = 31), or laparoscopic supracervical hysterectomy (n = 31).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women who are referred to the department
* benign condition requiring hysterectomy
* Dysmenorrohea/cyclic pelvic pain
* Informed consent

Exclusion Criteria:

* Women who are unable to communicate in Norwegian language.
* Women with a previous history of cervical dysplasia, with cellular changes suggestive of dysplasia in preoperative cervical smear.
* Women with atypical hyperplasia or malignancy in preoperative endometrial biopsy.
* Women with a substantially enlarged uterus requiring abdominal hysterectomy or not suitable for TLH (> 12 week amenorrhea).
* Women with a concomitant condition requiring uni- or bilateral oophorectomy.
* Postmenopausal women.
* Women with no dysmenorrohea/cyclic pelvic pain (<1 on a 10-point visual analogue scale).
* Women with deep infiltrating endometriosis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain reduction after the procedure. Occurrence and intensity of pelvic pain after the procedure. | 12 months after the procedure
  10-point visual analogue scale. Values are given as median (range), mean (sd) or n (%).

SECONDARY OUTCOMES:
Patient satisfaction after the procedure | 12 months after the procedure
  10-point visual analogue scale. Values are given as median (range) or mean (sd).
Occurrence of vaginal bleeding after the procedure | 12 months after the procedure
  Values are given as no bleeding, n (%); cyclical bleeding, n (%); irregular bleeding, n (%); bleeding related to sexual activity, n (%).
Improvement in patient Quality of Life after the procedure | 12 months after the procedure
  SF 36, Values are given as median (range) or mean (sd).
Frequency of perioperative and postoperative complications. | Perioperative and the periode 12 months after the prosedure
  Values are given as n (%) and eventual complications are specified. Major complications: Major haemorrhage (requiring transfusion), Haematoma requiring transfusion or surgical drainage, Bowel injury, Ureteric injury, Bladder injury, Pulmonary embolus, Major anaesthesia problems, Unintended laparotomy, Wound dehiscence Minor complications: Hemorrhage not requiring transfusion, Infection (chest, wound, pelvic, other; or fever >= 38 ºC on any single occasion), Hematoma (Spontaneous drainage), Deep vein thrombosis, Cervical stump problems, Minor anaesthesia problems, Others
Frequency of menopause | 12 months after surgery
  Values are given as n (%)and serum levels of ostradiol, FSH, LH, AMH
Frequency of adenomyosis in specimen from the operation. | postoperative
  Frequency of adenomyosis in specimen from the operation. Values are given as n (%).
Frequency and grade of genital prolapse | 60 and 120 months after procedure
  Frequency and grade of genital prolapse 60 and 120 months after procedure(POP-Q). Values are given as n (%) Type of prolapse is specified according to POP-Q Staging Criteria 0-IV and as cystocele, rectocele, enterocele, vault prolapse or combined prolapse.
Volume of uterine corpus preoperative, location and size of fibromas, Weight of the removed uterus/uterine corpus. | Pre- and perioperative
  Volume of the uterine corpus preoperative (cm3). Values are given as median (range) or mean (sd). Size and location of fibromas preoperative (cm). Values are given as median (range) or mean (sd), and is specified by location. Weight of the removed uterus/uterine corpus (g). Values are given as median (range) or mean (sd).

CONTACTS AND LOCATIONS:
Overall Officials: Marit Lieng, MD PHD, Study Director — Dept. of Gynecology, Oslo University Hospital, Norway
Locations (1):
- Dept. of Gynecology, Oslo University Hospital, Oslo, Oslo County, Norway

REFERENCES:
- See also: Homepage of Oslo University Hospital — http://www.oslo-universitetssykehus.no